CLINICAL TRIAL: NCT06478446
Title: The Mediating Role of Death Anxiety in the Relationship Between Religious Attitudes and Spiritual Care Needs in Hemodialysis Patients: A Sample of Turkey
Brief Title: The Mediating Role of Death Anxiety in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Rukiye Burucu, Associate prof., Necmettin Erbakan University
Other Study IDs: NECMETTİN EU-
Record Dates: First submitted 2024-06-22; First posted 2024-06-27 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Hemodialysis Complication; Death Anxiety; Religious Stigmata
Keywords: Death anxiety; Hemodialysis; Religious attitudes; Renal failure; Spiritual Care Needs
MeSH Terms: conditions — Necrophobia; Renal Insufficiency | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — HD patients were observed and evaluated with three scales.

SUMMARY:
This study aimed to determine the mediating role of death anxiety in the relationship between religious attitudes and spiritual care needs of hemodialysis (HD) patients in Turkey. The research was designed as a descriptive and cross-sectional study. A total of 203 patients were included in the study. Descriptive Characteristics Form, Religious Attitude Scale (RAS), Spiritual Care Needs Scale (SCNS), and Death Anxiety Scale (DAS) were used for data collection. In this study, it was found that the indirect effect of religious attitudes on spiritual care needs was significant, and death anxiety mediated the relationship between religious attitudes and spiritual care needs (b= -1.754, 95% CI [-2.95, -0.65]). It can be concluded that death anxiety in HD patients directs individuals towards religious attitudes, and in this case, the need for spiritual care increases. In other words, death anxiety mediates the relationship between religious attitudes and spiritual care needs. Therefore, nurses should include spiritual care when providing nursing care for HD patients.

DETAILED DESCRIPTION:
Materials and Methods The research was designed as a descriptive and cross-sectional study. Population and Sample The population of the study consisted of patients undergoing hemodialysis treatment at Necmettin Erbakan University Medical Faculty Hospital.

Sample The data of Burucu and Cantekin (2022) were used to determine the sample size. In this study, it was reported that death anxiety in dialysis patients varied according to the type of dialysis. In the mentioned study, R2 was 0.062. According to the multiple regression results on death anxiety, it was determined that the study should be completed with at least 149 participants to achieve 80% power and an effect size of 0.066. According to Dunson and Bollen, Structural Equation Modeling can be adequately performed with small sample sizes (approximately 100). However, it is recommended that the sample size should be 200 or more. Therefore, the calculated number was increased by 35% in line with the literature and the sample size of the study was determined as 201. A total of 203 patients were included in the study.

Data Collection Tools Descriptive Characteristics Form, Religious Attitude Scale (RAS), Spiritual Care Needs Scale (SCNS), and Death Anxiety Scale (DAS) were used for data collection.

Data were collected face-to-face by the researchers in the hemodialysis (HD) unit. During data collection, protective measures were taken to prevent the risk of infection. The patients were informed about the study and their consent was obtained.

Ethical approval was obtained from the XXX University Health Sciences Scientific Research Ethics Committee, and necessary permissions were obtained from XXX University Medical Faculty Hospital. All stages of the study were completed in accordance with the STROBE checklist and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Being eighteen years of age or older
* Being a resident in Turkey
* To be continuing HD treatment
* Not having communication barriers

Exclusion Criteria:

* Non-Muslim individuals,
* Those who are in the last stage of the disease,
* Those undergoing cancer treatment
* Those with cognitive impairment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The data of Burucu and Cantekin (2022) were used to determine the sample size. In this study, it was reported that death anxiety in dialysis patients varied according to the type of dialysis. In the mentioned study, R2 was 0.062 (Burucu & Cantekin, 2023). According to the multiple regression results on death anxiety, it was determined that the study should be completed with at least 149 participants to achieve 80% power and an effect size of 0.066. According to Dunson and Bollen, Structural Equation Modeling can be adequately performed with small sample sizes (approximately 100) (Palomo, Dunson, & Bollen, 2007). However, it is recommended that the sample size should be 200 or more (Şen & Yılmaz, 2013). Therefore, the calculated number was increased by 35% in line with the literature (Yıldırım Kaptanoğlu, 2013) and the sample size of the study was determined as 201. A total of 203 patients were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
The mediating role of death anxiety on the impact of religious attitudes on spiritual care needs | 2.10.2023/30.02.2024
  It was evaluated whether there is a mediating role of death anxiety on the effect of religious attitudes on spiritual care needs

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided